CLINICAL TRIAL: NCT04944953
Title: Double-blinded, Randomized, Active Control, Single Center-designed, Phase I Clinical Trial to Evaluate the Safety and Efficacy for Improvement of Glabellar Lines of "HG-102" Compared to Botox® in Subjects With Moderate to Severe Glabellar Lines
Brief Title: To Compare the Safety and Efficacy of "HG-102" With Botox® in the Improvement of Moderate to Severe Glabellar Lines.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hugel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HG-BOT102GL-PI-01
Record Dates: First submitted 2021-06-11; First posted 2021-06-30 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Glabellar Lines
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Botulinum toxin type A(Botox®) (Active Comparator): Botulinum toxin type A(Botox®) 100 Unit
  Interventions: Drug: Botulinum Toxin Type A Injection [Botox]
- Botulinum toxin type A(HG-102) (Experimental): Botulinum toxin type A(HG-102) 100 Unit
  Interventions: Drug: Botulinum toxin type A injection [HG-102]

INTERVENTIONS:
Drug: Botulinum Toxin Type A Injection [Botox] — Single administration, Day 0, 20 units
  Other Names: Botox®
  Arms: Botulinum toxin type A(Botox®)
Drug: Botulinum toxin type A injection [HG-102] — Single administration, Day 0, 20 units
  Other Names: HG-102
  Arms: Botulinum toxin type A(HG-102)

SUMMARY:
To compare the safety and efficacy of "HG-102" with Botox® in the improvement of moderate to severe glabellar lines.

DETAILED DESCRIPTION:
Double-blinded, Randomized, Active control, Single center-designed, Phase I clinical trial to evaluate the safety and efficacy for improvement of Glabellar Lines of "HG-102" compared to Botox® in subjects with moderate to severe Glabellar Lines

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 19 and 65 at screening visit.
* Patients who voluntarily sign the informed consent.
* Patients who can comply with the study procedures and visit schedule.

Exclusion Criteria:

* Patients with infection, skin disorders, or scars at the glabellar region.
* Patients with facial palsy or the symptoms of blepharoptosis.
* Fertile women and men who have plans to conceive during pregnancy, breastfeeding and clinical trials or who do not agree to appropriate contraception.
* Subjects who are not eligible for this study based on investigator's judgement.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2021-09-02 (Actual); Study Completion 2021-12-16 (Actual)

PRIMARY OUTCOMES:
Adverse event and adverse drug reaction incidence rates | Baseline to week 16
Clinically-relevant changes in vital signs, physical exam, and laboratory testing assessed by medical personnel | 16 weeks (during the clinical trial)

SECONDARY OUTCOMES:
Responder rate of improvement in glabellar lines with Physician's rating line severity | Baseline to week 4, 8, 12, 16
  Improvement rate of glabellar lines at maximum frown with Physician's rating line severity at 4, 8, 12, 16 weeks post injection
Responder rate of improvement in glabellar lines with investigator's photo assessment | Baseline to week 4, 8, 12, 16
  Improvement rate of glabellar lines at maximum frown with investigator's photo assessment at 4, 8, 12, 16 weeks post injection
Responder rate of improvement in glabellar lines with Physician's rating line severity | Baseline to week 4, 8, 12, 16
  Improvement rate of glabellar lines at rest with Physician's rating line severity at 4, 8, 12, 16 weeks post injection
Responder rate of improvement in glabellar lines with investigator's photo assessment | Baseline to week 4, 8, 12, 16
  Improvement rate of glabellar lines at rest with investigator's photo assessment at 4, 8, 12, 16 weeks post injection
Changes in grade by physician's rating line severity for glabellar lines | Baseline to week 4, 8, 12, 16
  Changes in grade(range from 0(None) to 3(Severe)) by physician's rating line severity for glabellar lines at each visit compared to baseline
Responder rate of improvement in glabellar lines with Subject's improvement assessment | Baseline to week 4, 8, 12, 16
  Improvement rate of glabellar lines with Subject's improvement assessment at 4, 8, 12, 16 weeks post injection
Subject's satisfaction rate | Baseline to week 4, 8, 12, 16
  Subject's satisfaction rate of improvement in glabellar lines at 4, 8, 12, 16 weeks post injection
The severity of pain evaluated by the subject's Simple Descriptive Scale (SDS) | Baseline
  The severity of pain evaluated by the subject's Simple Descriptive Scale (SDS) at immediately and about 30 minutes post injection (severity range is from 1(no pain) to 5(unbearable pain))

CONTACTS AND LOCATIONS:
Locations (1):
- Konkuk University Medical Center, Seoul, Korea, South Korea